CLINICAL TRIAL: NCT02267356
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy and Safety of VT-1161 Oral Tablets in the Treatment of Patients With Distal Lateral Subungual Onychomycosis of the Toenail
Brief Title: A Study to Evaluate the Efficacy and Safety of Oral VT-1161 in Patients With Onychomycosis of the Toenail
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Viamet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: VMT-VT-1161-CL-005
Record Dates: First submitted 2014-10-08; First posted 2014-10-17 (Estimated); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — VT-1161

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Low dose 12-week (Experimental): 2 VT-1161 150mg tablets and 2 placebo tablets once daily for 2 weeks, then once weekly for 10 weeks, followed by 4 placebo tablets once weekly for 12 weeks
  Interventions: Drug: VT-1161
- Low dose 24-week (Experimental): 2 VT-1161 150mg tablets and 2 placebo tablets once daily for 2 weeks, then once weekly for 22 weeks
  Interventions: Drug: VT-1161
- High dose 12-week (Experimental): 4 VT-1161 150mg tablets once daily for 2 weeks, then once weekly for 10 weeks, followed by 4 placebo tablets once weekly for 12 weeks
  Interventions: Drug: VT-1161
- High dose 24-week (Experimental): 4 VT-1161 150mg tablets once daily for 2 weeks, then once weekly for 22 weeks
  Interventions: Drug: VT-1161
- Placebo (Placebo Comparator): 4 placebo tablets once daily for 2 weeks, then once weekly for 22 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VT-1161
  Arms: High dose 12-week; High dose 24-week; Low dose 12-week; Low dose 24-week
Drug: Placebo
  Arms: Placebo

SUMMARY:
Several properties of VT-1161 suggest that it might be a safer and more effective treatment for onychomycosis of the toenail (also known as toenail fungus) than other oral antifungal medicines.

This study will evaluate the effectiveness and safety of VT-1161 for the treatment of toenail onychomycosis and consists of a screening phase, a 24-week treatment phase in which the patient will take either active drug, placebo or a combination of the 2 (according to random assignment), an initial observational phase of 36 weeks and an additional observational study extension of 9 months.

The additional 9-month observational study extension was added with a protocol amendment and patient participation was optional.

ELIGIBILITY:
Key Inclusion Criteria:

Distal subungual onychomycosis of the great toenail, affecting at least ≥25 to ≤75% of nail.

Positive culture for dermatophytes and positive KOH.

Nail ≤ 3 mm thick at the distal end.

At least ≥ 2 mm of the proximal end of the great toenail must be free of infection.

Subjects must be able to swallow tablets.

Women of childbearing potential and males must use acceptable birth control methods throughout the study.

Key Exclusion Criteria:

Presence of subungual hematoma or melanonychia.

Presence of dermatophytoma/nail streaks and severe onychorrhexis.

Significant dystrophy or anatomic abnormalities of the great toenail.

Presence of any other infections of the foot.

Evidence of clinically significant major organ disease.

Poorly controlled diabetes mellitus.

Onychomycosis involving more than 8 toe nails.

Recent use of systemic antifungal therapy.

Recent of any topical antifungal nail therapy.

Recent use of systemic corticosteroid therapy.

Recent use of immunosuppressive medication.

History of prolonged QT intervals.

Known human immunodeficiency virus (HIV) infection.

Known significant renal or hepatic impairment.

Known history of intolerance or hypersensitivity to azole antifungal drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2016-10-18 (Actual); Study Completion 2017-07-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - The Kirklin Clinic of UAB Hospital, Birmingham, Alabama
  - Radiant Research, Tucson, Arizona
  - Dermatology Specialists, Inc, Oceanside, California
  - Therapeutics Clinical Research, San Diego, California
  - Center For Clinical Research, San Francisco, California
  - Radiant Research, Santa Rosa, California
  - International Dermatology Research, Miami, Florida
  - Radiant Research, Pinellas Park, Florida
  - Northwest Clinical Trials, Boise, Idaho
  - Gateway Health Center, Newburgh, Indiana
  - Mid Atlantic Research Center for Health, Baltimore, Maryland
  - Associated Skin Care Specialist Minnesota Clinical Study Center, Minneapolis, Minnesota
  - Skin Specialists, PC, Omaha, Nebraska
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Forest Hills Dermatology Group, Forest Hills, New York
  - Skin Search of Rochester, Rochester, New York
  - Radiant Research, Akron, Ohio
  - Radiant Research, Cincinnati, Ohio
  - Radiant Research, Columbus, Ohio
  - Oregon Dermatology & Research Center, Portland, Oregon
  - Oregon Medical Research Center, Portland, Oregon
  - Paddington Testing Company, Philadelphia, Pennsylvania
  - Martin Foot and Ankle, York, Pennsylvania
  - Radiant Research, Greer, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - The Skin Wellness Center, Knoxville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch, Austin, Texas
  - J&S Clinical Studies, College Station, Texas
  - Ashton Podiatry Associates, PA, Dallas, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - The Education And Research Foundation, Inc., Lynchburg, Virginia
  - Virginia Clinical Research, Inc., Norfolk, Virginia

REFERENCES:
- [Derived] Elewski B, Brand S, Degenhardt T, Curelop S, Pollak R, Schotzinger R, Tavakkol A. A phase II, randomized, double-blind, placebo-controlled, dose-ranging study to evaluate the efficacy and safety of VT-1161 oral tablets in the treatment of patients with distal and lateral subungual onychomycosis of the toenail. Br J Dermatol. 2021 Feb;184(2):270-280. doi: 10.1111/bjd.19224. Epub 2020 Jul 13. PMID 32421854

RESULTS

PARTICIPANT FLOW:
Period: Initial Study
Arm/Group | Low Dose 12-week | Low Dose 24-week | High Dose 12-week | High Dose 24-week | Placebo
Started | 53 | 53 | 52 | 54 | 47
Completed | 47 | 48 | 42 | 43 | 42
Not Completed | 6 | 5 | 10 | 11 | 5
Period: Study Extension
Arm/Group | Low Dose 12-week | Low Dose 24-week | High Dose 12-week | High Dose 24-week | Placebo
Started (Not all subjects completing initial study continued in study extension. Continuation was optional.) | 33 | 37 | 30 | 32 | 26
Completed | 32 | 37 | 29 | 30 | 26
Not Completed | 1 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population data is for initial 60-week study only.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose 12-week | Low Dose 24-week | High Dose 12-week | High Dose 24-week | Placebo | Total
Number analyzed (Participants) | 53 | 53 | 52 | 54 | 47 | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (9.41) | 50.4 (10.28) | 49.4 (12.79) | 49.0 (10.45) | 52.7 (11.69) | 50.0 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 13 | 9 | 9 | 51
  Male | 41 | 45 | 39 | 45 | 38 | 208

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects in the Intent-to-treat Population With Complete Cure, Defined as Clinical AND Mycological Cure, at Week 48
Description: Complete cure was defined as 0% nail involvement and an Investigator Global Assessment (IGA) score of 0. Mycological cure was defined as negative potassium hydroxide (KOH) and negative dermatophyte culture.
  Investigator Global Assessment (IGA) scoring:
  0: 0% nail involvement
  1. >0% to ≤10% nail involvement
  2. >10% to <25% nail involvement
  3. ≥25% to ≤50% nail involvement
  4. >50% to ≤75% nail involvement
  5. >75% nail involvement
Time Frame: 48 weeks
Population: Initial 60-week study data. Study extension data not applicable.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose 12-week | Low Dose 24-week | High Dose 12-week | High Dose 24-week | Placebo
Number analyzed (Participants) | 53 | 53 | 52 | 54 | 47
Participants | 17 | 19 | 22 | 18 | 0

2. Primary Outcome: Study Extension - Number of Subjects Who Experienced Treatment-emergent Adverse Events and Lab Abnormalities
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose 12-week | Low Dose 24-week | High Dose 12-week | High Dose 24-week | Placebo
Number analyzed (Participants) | 33 | 37 | 30 | 32 | 26
Participants | 8 | 5 | 7 | 9 | 6

ADVERSE EVENTS:
Description: Reported non-serious adverse event data do not include events reported during the study extension. No serious adverse events were reported during the study extension. 35 subjects experienced non-serious adverse events, as follows:
  Low-dose 12-week: 8 subjects; Low-dose 24-week: 5 subjects; High-dose 12-week: 7 subjects; High-dose 24-week: 9 subjects; Placebo: 6 subjects.
Groups:
- Low Dose 12-week: Loading doses of VT-1161 300mg once daily for 2 weeks, then 300mg once weekly for 10 weeks, followed by placebo for 12 weeks
- Low Dose 24-week: Loading doses of VT-1161 300mg once daily for 2 weeks, then 300mg once weekly for 22 weeks
- High Dose 12-week: Loading doses of VT-1161 600mg once daily for 2 weeks, then 600mg once weekly for 10 weeks, followed by placebo for 12 weeks
- High Dose 24-week: Loading doses of VT-1161 600mg once daily for 2 weeks, then 600mg once weekly for 22 weeks
- Placebo: Matching placebo tablets for 24 weeks
Arm/Group | Low Dose 12-week | Low Dose 24-week | High Dose 12-week | High Dose 24-week | Placebo
Serious Adverse Events (participants affected / at risk) | 1/53 | 1/53 | 2/52 | 5/54 | 2/47
Other Adverse Events (participants affected / at risk) | 29/53 | 26/53 | 31/52 | 36/54 | 26/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose 12-week (N=53) | Low Dose 24-week (N=53) | High Dose 12-week (N=52) | High Dose 24-week (N=54) | Placebo (N=47)
Hemorrhagic anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Postmenopausal hemmorage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Artery dissection (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose 12-week (N=53) | Low Dose 24-week (N=53) | High Dose 12-week (N=52) | High Dose 24-week (N=54) | Placebo (N=47)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Congenital aural fistula (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2 | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0
Meibomian gland dysfunction (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 2
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 4 | 4 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 0
Edema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 1 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 5 | 0 | 4 | 2 | 2
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 4 | 4 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 5 | 5 | 4
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Nail injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Tooth avulsion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Traumatic hematoma (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 1 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 1 | 0
Blood testosterone decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Electrocardiogram change (Investigations) | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 1 | 0
Bunion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
7th nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 3 | 0
Dyskinesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 1 | 0 | 1
Hyperesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 3 | 2 | 5 | 3 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Scar (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 1 | 0 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither Institution nor Principal Investigator shall publish the results of the Trial without the prior written consent of Sponsor, which it may withhold in its sole discretion.